CLINICAL TRIAL: NCT07207928
Title: Evaluation of Clinical Outcomes, Tolerability, and Costs of Avelumab as First-Line Maintenance Therapy and Pembrolizumab as Second-Line Therapy in Patients With Advanced Urothelial Cancer Without Disease Progression After First-Line Platinum-Based Chemotherapy: A Multicenter Retro-Prospective Observational Study in Real-World Clinical Practice
Brief Title: Evaluation of Clinical Outcomes, Tolerability, and Costs of Avelumab Maintenance and Pembrolizumab Second-Line Therapy in Advanced Urothelial Cancer.
Acronym: AvePem
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: Ospedale Mater Salutis-Legnago(Verona), Italy (Unknown); Casa di Cura Dott. Pederzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 339CET
Record Dates: First submitted 2025-09-08; First posted 2025-10-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Urothelial Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate the clinical outcomes, side effects, and costs of Avelumab maintenance therapy in first-line and Pembrolizumab in second-line for platinum-fit patients with advanced urothelial cancer who have not shown disease progression after 4-6 cycles of platinum-based first-line chemotherapy.

Researchers will compare the effects of Avelumab (used as maintenance in first-line) and Pembrolizumab (used in second-line) to see if there are differences in clinical outcomes, toxicity profiles, and costs.

Participants will:

Receive Avelumab as maintenance therapy in the first-line or Pembrolizumab in the second-line as per standard clinical practice.

Be monitored for clinical outcomes, side effects, and costs over a period of up to 12 months prospectively and 10 years retrospectively.

DETAILED DESCRIPTION:
Retrospective-prospective study

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* ECOG PS 0-2
* Diagnosis of pathologically confirmed stage IV urothelial cancer, regardless of PD-L1 status
* Patients treated with platinum-based chemotherapy (Cisplatin or Carboplatin) in the first-line setting who have not shown disease progression after 4-6 cycles of chemotherapy
* Patients receiving Avelumab as maintenance therapy in the first-line setting or Pembrolizumab in the second-line setting
* Availability of hospital and/or outpatient medical records for clinical data collection
* Ability to understand and willingness to provide informed consent, or deceased patients at the time of enrollment, in compliance with Article 110 of the Privacy Code and the safeguards established by the Data Protection Authority in Provision No. 298 of May 9, 2024.

Exclusion Criteria:

* History of another malignancy or concurrent malignancy (except for cured non-melanoma skin cancer, low-risk prostate cancer, T1/T2 glottic cancer, stage 0 or I breast cancer, non-invasive bladder cancer, or in situ cervical cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced urothelial cancer without disease progression after 4-6 cycles of first-line platinum-based chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 1 year
  Radiologic Progression-Free Survival (PFS) Evaluation in patients with advanced platinum-fit urothelial carcinoma who have no disease progression after 4-6 cycles of first-line platinum-based chemotherapy. These patients are treated with Avelumab in first-line maintenance therapy, or Pembrolizumab in second-line therapy. Radiologic progression is defined as the time from the start of first-line platinum-based chemotherapy to the date of radiologic progression (according to RECIST v1.1) after initiation of Avelumab maintenance therapy in the first-line or Pembrolizumab in the second-line, or death from any cause.
Overall Survival | 1 year
  Overall Survival (OS) Evaluation in patients with advanced platinum-fit urothelial carcinoma who have no disease progression after 4-6 cycles of first-line platinum-based chemotherapy. These patients are treated with Avelumab in first-line maintenance therapy, or Pembrolizumab in second-line therapy.

SECONDARY OUTCOMES:
Duration of Subsequent Oncologic Treatments | 1 year
  Duration of Subsequent Oncologic Treatments in patients with advanced platinum-fit urothelial carcinoma who have no disease progression after 4-6 cycles of first-line platinum-based chemotherapy treated with Avelumab in first-line maintenance therapy compared to patients treated with Pembrolizumab in second-line therapy.
Adverse Events | 1 year
  Adverse Events of Any Grade Related to Treatment according to CTCAE 5.0, in patients with advanced platinum-fit urothelial carcinoma who have no disease progression after 4-6 cycles of first-line platinum-based chemotherapy treated with Avelumab in first-line maintenance therapy, compared to patients treated with Pembrolizumab in second-line therapy. Adverse events will be evaluated based on their severity and relationship to the treatment received.
Serious Adverse Events | 1 year
  Adverse Events of Grade 3 or Higher Related to Treatment according to CTCAE 5.0, in patients with advanced platinum-fit urothelial carcinoma who have no disease progression after 4-6 cycles of first-line platinum-based chemotherapy. These patients are treated with Avelumab in first-line maintenance therapy, compared to patients treated with Pembrolizumab in second-line therapy. Adverse events of grade 3 or higher will be monitored and assessed for their relationship to the treatment received.
Overall Cost of Oncologic Therapy | 1 year
  Overall Cost of Oncologic Therapy in patients with advanced platinum-fit urothelial carcinoma who have no disease progression after 4-6 cycles of first-line platinum-based chemotherapy treated with Avelumab in first-line maintenance therapy, compared to patients treated with Pembrolizumab in second-line therapy. The cost will be evaluated for each treatment approach and compared between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Integrata di Verona, Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No